CLINICAL TRIAL: NCT07099131
Title: Effective Interventions to Overcome Severe Gag Reflex
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6213
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gagging
MeSH Terms: conditions — Gagging | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Unblinded. Subjects will be randomized. The three intervention groups are : Acupuncture (CV-24), Tape and Anesthetic Spray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Acupuncture (CV-24) (Experimental): A 6C file (endodontic instrumentation file) will be placed on the patient's mentolabial fold (CV24). This file will be concealed by a small paper cup; A clean alcohol wipe will be used to clean the mentolabial area prior to placing the "acupuncture needle" (6 C-File).
  Interventions: Device: Acupuncture
- Tape (Experimental): A piece of commercially available masking tape will be adhered to the patient's mentolabial fold and concealed by the small paper cup
  Interventions: Genetic: Masking Tape
- Anesthetic spray (Experimental): Will be applied to back of the throat for 10 seconds; their chin will also be concealed from the GSI examiner using a small cup and masking tape.
  Interventions: Drug: Anesthetic spray

INTERVENTIONS:
Drug: Anesthetic spray — will be applied to back of the throat for 10 seconds; their chin will also be concealed from the GSI examiner using a small cup and masking tape.
  Arms: Anesthetic spray
Device: Acupuncture — A 6C file (endodontic instrumentation file) will be placed on the patient's mentolabial fold (CV24). This file will be concealed by a small paper cup; A clean alcohol wipe will be used to clean the mentolabial area prior to placing the "acupuncture needle" (6 C-File).
  Arms: Acupuncture (CV-24)
Genetic: Masking Tape — A piece of commercially available masking tape will be adhered to the patient's mentolabial fold and concealed by the small paper cup
  Arms: Tape

SUMMARY:
The purpose of this study is to evaluate the use of various techniques in alleviating gag reflex following gag reflex stimulation.

Primary aim: To compare if there is any reduction in gag reflex from each of the following interventions

* Acupuncture (CV-24)
* Tape
* Anesthetic spray Secondary aim: to compare the degree of gag reduction

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of various techniques in alleviating gag reflex following gag reflex stimulation.

Primary aim: To compare if there is any reduction in gag reflex from each of the following interventions

* Acupuncture (CV-24)
* Tape
* Anesthetic spray Secondary aim: to compare the degree of gag reduction

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older (individuals below 18 years will be excluded from the study as the study procedures might not be well tolerated by them, and they are not the primary population on which these procedures are used).
* Students, faculty, or staff of Tufts SDM
* Subjects who score a 2 or higher on the Gagging Severity Index (GSI)7 and have a positive gag reflex response when stimulated with a cotton swab at the base of the tongue/uvula/tonsil region.

Exclusion Criteria:

* Adults unable to consent (cognitively impaired adults)
* Wards of the state
* Pregnant women (those that are self-reported)
* Current use of anticoagulants
* Allergy to xylocaine
* Those with bleeding disorders
* Those who participated in the Calibration phase of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2027-12-07 (Estimated); Study Completion 2028-12-07 (Estimated)

PRIMARY OUTCOMES:
Change in Gag Reflex Severity Index (GSI) Score From Pre- to Post-Intervention | 90 minutes per subject
  Change in Gag Reflex Severity Index (GSI) Score From Baseline to Post-Intervention
  * Acupuncture (CV-24)
  * Tape
  * Anesthetic spray
  Gag reflex severity will be assessed by clinicians using the Gagging Severity Index (GSI), based on definitions set by Dickinson and Fiske. GSI will first be recorded after initial gag stimulation with a cotton swab. Following randomization to one of three interventions (acupuncture, anesthetic spray, or masking tape), GSI will be recorded again. The change in GSI score will be used to measure change in gag response.

SECONDARY OUTCOMES:
Self-Reported Degree of Gag Reflex Reduction Using Visual Analog Scale (VAS) | Immediately post-intervention during single study visit
  Participants will complete an in-session survey to rate their gag reflex severity after the assigned intervention using a Visual Analog Scale (VAS). The VAS rating reflects the participant's perception of gag reduction following either acupuncture at CV24, anesthetic spray, or masking tape application.

CONTACTS AND LOCATIONS:
Overall Officials: Devon Ptak, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No